CLINICAL TRIAL: NCT06261905
Title: Exploration of Baseline Alterations on the Dopamine D2/D3 Receptor System and the Effects of Vitamin D in Opioid Use Disorder: an [11C]-PHNO Study
Brief Title: Vitamin D in OUD: Exploration of Alterations on the Dopamine D2/D3 Receptor System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2000036908; 000 (Other: CTGTY)
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: Vitamin D
MeSH Terms: conditions — Opioid-Related Disorders | interventions — naxagolide; Calcitriol; Vitamin D; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: This is primarily a within-subject, two scan, randomized, double-blind, placebo-controlled study design. Healthy control subjects will only complete one scan to serve as a baseline comparison for subjects with OUD.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcitriol (Active Comparator): Subjects with OUD will receive a baseline MRI. On the night before and day of testing, subjects with OUD will receive two doses of calcitriol (3.0mcg total), followed by PHNO injection and PET Scan for the calcitriol condition. All subjects will complete the study with both active calcitriol and a placebo control and the order these interventions are received will be randomized.
  Interventions: Drug: [11C]-PHNO; Dietary Supplement: Calcitriol; Procedure: PET Scan
- Placebo (Placebo Comparator): Subjects with OUD will receive a baseline MRI. On the night before and day of testing, subjects with OUD will receive two doses of an inactive placebo, followed by PHNO injection and PET Scan for the placebo condition. All subjects will complete the study with both active calcitriol and a placebo control and the order these interventions are received will be randomized.
  Interventions: Drug: [11C]-PHNO; Other: Placebo Control; Procedure: PET Scan

INTERVENTIONS:
Drug: [11C]-PHNO — PHNO is used as a tracer for in-vivo imaging.
  Other Names: PHNO
Dietary Supplement: Calcitriol — Calcitriol is an active form of Vitamin D and is given in 3 0.5mcg capsules per dose.
  Other Names: Vitamin D
  Arms: Calcitriol
Other: Placebo Control — A placebo is an inert capsule, which contains no active ingredients. The placebo will be given in 3 0.5mcg capsules per dose.
  Arms: Placebo
Procedure: PET Scan — A high resolution PET Scan performed using a NeurExplorer CT scanner.

SUMMARY:
The research team is investigating Opioid Use Disorder (OUD), a disorder characterized by dysregulated dopaminergic tone, to evaluate the mechanisms of adjunctive treatment with calcitriol. The investigators will recruit 12 subjects with OUD and 12 healthy subjects to participate in a double-blind, randomized study design where subjects will complete up to 2 Positron Emission Tomography (PET) scans using [11C]-PHNO. The investigators will compare subjects in differences between their own study days and in differences between healthy control subjects and subjects with OUD.

DETAILED DESCRIPTION:
Previous research has indicated that Dopamine (DA) may play a role in withdrawal and dependence in Opioid Use Disorder (OUD). The present study will investigate dopamine receptor availability in 12 subjects with OUD compared with 12 HC subjects using [11C](+)-PHNO and the impact of calcitriol on these receptors.

Research has indicated that a common feature in substance use disorders (SUD) is a hypo-dopaminergic state. Further, preclinical and observational research has pointed to a possible benefit of calcitriol in individuals who have OUD and our research group has previously shown the potential benefits of calcitriol on addressing this hypo-dopaminergic state. If successful, the results of this research study may improve the standard treatment for OUD through calcitriol supplementation.

Specifically, the present study seeks to address the following aims:

Specific Aim 1: As part of a between-subject study design, to determine whether acute calcitriol (vs. placebo) administration is associated with greater dopamine (DA) release in the caudate, putamen, ventral striatum (VST), and substantia nigra / ventral tegmental area (SN/VTA) of subjects with OUD compared to healthy control subjects (HCs).

Specific Aim 2: As part of a within-subject, two-day study design, to determine whether acute calcitriol (vs. placebo) administration is associated with greater dopamine (DA) release in the caudate, putamen, ventral striatum (VST), and substantia nigra / ventral tegmental area (SN/VTA) of subjects with OUD.

Specific Aim 3: To determine whether acute calcitriol (vs. placebo) administration is associated with higher spontaneous eyeblink rate, a non-PET indicator of higher dopamine activity, among subjects with OUD.

Specific Aim 4: To determine whether acute calcitriol (vs. placebo) administration is associated with better performance on neurocognitive measures (e.g., the Continuous Performance Task or CPT-IP and the Probabilistic Reversal Learning Task or PRLT) among subjects with OUD.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years
2. Voluntary, written, informed consent
3. Physically healthy by medical history, physical, neurological, ECG, and laboratory examinations
4. Meets the criteria for OUD, as determined by the Structured Clinical Interview for DSM-5 (SCID)
5. Stable and receiving buprenorphine treatment for OUD
6. For females, non-lactating, with a negative serum or urine pregnancy (hCG) test
7. Lab results without clinically relevant findings (e.g., renal function, electrolytes, and vitamin D levels)
8. English speaking

Exclusion criteria:

1. Medical contraindication to calcitriol administration (e.g., history of hypersensitivity to calcitriol or any component of the formulation, hypercalcemia or vitamin D toxicity)
2. History of substance dependence (e.g., alcohol, sedative hypnotics), except for nicotine and opiates.
3. A primary major DSM-5 psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) as determined by the SCID, except for Opioid Use Disorder and related conditions.
4. A history of significant medical (e.g., cardiovascular, diabetic/metabolic) or neurological (e.g., cerebrovascular accidents, seizure, traumatic brain injury) illness
5. Positive answers on the cardiac history questionnaire that may place the subject at higher risk, as determined by the study physician's review of both the questionnaire responses and screening ECG. If there is concern for the subject's safety due to these assessments, research staff will consult a Yale PET Center affiliated cardiologist prior to including the subject for the study.
6. Current use of psychotropic and/or potentially psychoactive prescription medications
7. Receiving medications for OUD other than buprenorphine (e.g., methadone treatment)
8. For females, laboratory (β-HCG) or physical evidence of pregnancy/lactation
9. MRI-incompatible implants and other contraindications for MRI (i.e., aneurysm clip, metal fragments, internal electrical devices such as a cochlear implant, spinal cord stimulator or pacemaker)
10. History of claustrophobia or feeling of inability to lie still on his/her back for the PET or MRI scans
11. History of any bleeding disorder or current anticoagulant therapy
12. Donation or loss of 550 mL of blood or more (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to the first test day.
13. Use of any prescription medications and/or over-the-counter medications, vitamins and/or herbal supplements which could have a negative clinical interaction with calcitriol or which could confound scientific results of the study, within 2 weeks prior to each test day (e.g., thiazide diuretics, Mg based antiacids, digoxin, etc,).
14. Serum levels of 25(OH)D3 below 12 ng/ml.
15. Morbid obesity i.e., BMI over 35 (more prone to lower vitamin D levels)
16. Subjects with history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year.
17. Subjects with current, past or anticipated exposure to radiation in the workplace
18. History of kidney stones within the past 5 years
19. Any degree of renal failure
20. History of parathyroid disorder (hyper or hypoparathyroidism)
21. History of osteoporosis or any pathologic fractures
22. Vitamin D supplementation in any form in the past 3 months
23. Known hypersensitivity to [11C]-PHNO or calcitriol
24. Malabsorption syndromes (i.e., Celiac sprue)
25. Serum corrected calcium > 10.5 mg/dl or phosphate > 4.2 mg/dL

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Non-displaceable Tracer Binding Potentials (BPND) | One 120-minute scan.
  BPND is a metric that assesses the level of dopamine activity in a priori regions of interest. For Specific Aim 1, the investigators plan to assess the differences in baseline BPND in dopamine D2/D3 receptors between healthy control subjects and the baseline placebo-controlled scan for subjects with OUD.
Non-displaceable Tracer Binding Potentials (BPND) | Two 120-minute scans, at least 6 days apart between study conditions.
  BPND is a metric that assesses the level of dopamine activity in a priori regions of interest. For Specific Aim 2, the investigators plan to assess the differences in BPND in dopamine D2/D3 receptors within subjects who have OUD. The investigators will compare BPND on the placebo-controlled experimental day and BPND on the active calcitriol experimental day.

SECONDARY OUTCOMES:
Spontaneous Blink Rate (SBR) | Two 5-minute tasks, at least 6 days apart between study conditions.
  SBR is a metric that may assess levels of dopamine activity, without requiring the subject to undergo a PET scan. Subjects will be recorded for approximately 5 minutes to assess blink rate during each experimental day to address Specific Aim 3.
Continuous Performance Task - Identical Pairs (CPT-IP) | Two 10-minute tasks, at least 6 days apart between study conditions.
  The CPT-IP is a computer based test where subjects are shown a random sequence of numbers (2-digit, 3-digit, and 4-digit) and are instructed to press a button as quickly and accurately as possible with their preferred hand when a number repeats. Subjects are instructed to withhold their response for any other sequence of numbers. Subjects will complete this task on each experimental day to address Specific Aim 4.
Probabilistic Reversal Learning Task (PRLT) | Two 10-minute tasks, at least 6 days apart between study conditions.
  The PRLT is a computer based test where subjects are instructed to select a card from three randomly sorted piles and are asked to try to maximize their score in the task. Subjects will complete this task on each experimental day to address Specific Aim 4.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States